CLINICAL TRIAL: NCT00935870
Title: Bioactive Glass (S53P4) as Bone Graft Substitute in Operative Treatment of Depressed Lateral Condyle Fractures, Benign Bone Tumour Cavities and in Spinal Fusion - a 10 Years Follow-up and Bone Density Study.
Brief Title: Bioactive Glass as Bone Graft Substitute in Operative Treatment of Bone - a 10 Years Follow-up Study
Status: Completed | Type: Observational
Sponsor: Vivoxid Ltd (Industry)
Responsible Party: Kirsi Rosenqvist, Clinical Research Manager, Vivoxid Ltd
Other Study IDs: 1005-3
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Depressed Lateral Condyle Fracture; Benign Bone Tumour Cavity; Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: DEPRESSED LATERAL CONDYLE FRACTURE
  Interventions: Device: Bioactive glass and/or autogenous bone
- B: BENIGN BONE TUMOR
  Interventions: Device: Bioactive glass and/or autogenous bone
- C: SPINAL FUSION
  Interventions: Device: Bioactive glass and/or autogenous bone

INTERVENTIONS:
Device: Bioactive glass and/or autogenous bone — No intervention in the current study (10-year follow-up study)

SUMMARY:
The main aim is to evaluate the long-term safety and bone healing in the operated area and to compare bioactive glass granules with autogenous bone as a filler material.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained; Participation of previous clinical investigation with bioactive glass

Exclusion Criteria:

* The subject is unlikely to adhere to study procedures
* Concurrent disease or condition that in the opinion of the investigator is contraindicating participation
* Simultaneous participation in another medical device or investigational drug trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated to previous clinical investigations with bioactive glass about 10 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lindfors, MD, Principal Investigator — Turku University Hospital/Helsinki University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland